CLINICAL TRIAL: NCT00896974
Title: A Pilot Study of the Novel Retinoid, 9cUAB30 to Determine Preliminary Pharmacokinetics
Brief Title: Study of 9cUAB30 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00907; NCI-2009-00907 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CO06901; CDR0000610174; WCCC-CO06901 (Other: University of Wisconsin Hospital and Clinics); UWI06-8-03 (Other: DCP); N01CN35153 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2014-02

CONDITIONS: No Evidence of Disease
MeSH Terms: interventions — UAB 30

ARMS (1):
- Arm I (Experimental): Participants receive a single dose of oral 9cUAB30 on day 1.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Retinoid 9cUAB30

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Retinoid 9cUAB30 — Given orally
  Other Names: 9cUAB30

SUMMARY:
This research study is looking at 9cUAB30 in healthy participants. Studying samples of blood and urine from healthy participants may help doctors learn more about how 9cUAB30 is used by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the single-dose pharmacokinetics of 9cUAB30 in healthy volunteers.

SECONDARY OBJECTIVES:

I. To determine the toxicities of this drug in these participants. II. To correlate the pharmacokinetics with the toxicity of this drug in these participants.

OUTLINE:

Participants receive a single dose of oral 9cUAB30 on day 1. Blood and urine samples are collected at baseline, periodically on day 1, and then on day 8 for pharmacokinetic studies by high performance liquid chromatography.

After completion of treatment, participants are followed at days 8 and 30.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Karnofsky performance status (PS) 70-100% (ECOG PS 0-1)
* WBC ≥ 3,000/mm³
* Platelet count ≥ 100,000mm³
* Hemoglobin > 10 g/dL
* Bilirubin ≤ 1.4 mg/dL
* AST ≤ 1.5 times normal
* Creatinine normal
* Sodium 135-144 mmol/L
* Potassium 3.2-4.8 mmol/L
* Chloride 85-114 mmol/L
* Bicarbonate > 11 mEQ/dL
* Fasting triglycerides ≤ 1.5 times upper limit of normal (ULN)
* Fasting cholesterol ≤ 1.5 times ULN
* Not pregnant or nursing

  * No nursing during and for 30 days after completion of study treatment
* Negative pregnancy test
* Fertile participants must use effective contraception prior to, during, and for 1 month after completion of study treatment

  * No low-dose progesterone only birth control pills
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatricillness or social situation that would limit compliance with study requirements
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to retinoids
* No other concurrent investigational agents
* No concurrent lipid-lowering agents
* No concurrent medications that may interact with 9cUAB30 (e.g., St.John's wort, ketoconazole, vitamin A, tetracycline, or oral corticosteroids)
* No other concurrent topical or oral retinoids (e.g., retinol, retinal, tretinoin [Retin-A], isotretinoin, alitretinoin, etretinate, acitretin,tazarotene, or bexarotene)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Single dose pharmacokinetics of 9cUAB30 | 0, 30, 45, 60, and 90 minutes, 2, 4, 6, 8, 12, 16, 18, 20, and 24 hours, and day 8
  Scatterplots will be used to explore possible associations. Jonckheere-Terpstra trend test will be performed to determine the significance of the association between increasing dose level and each of the pharmacokinetic parameters. A Spearman rank correlation analysis will be performed to determine the relationship between actual dose administered and the pharmacokinetic parameters. Additionally, logistic regression analyses will be performed to correlate PK parameters with toxicity.

SECONDARY OUTCOMES:
Grade II or greater toxicities assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 30 days
  Patient toxicity will be summarized in several ways; the presence or absence of any toxicities, worst CTCAE grade, and strongest investigator-defined relationship will all be examined and characterized by dose. The different pharmacokinetic measures will be correlated with toxicity measures with polyserial correlation, a method for estimating the correlation between a continuous variable and an ordinal variable whose underlying distribution is continuous.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Bailey, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States